CLINICAL TRIAL: NCT02083731
Title: Mesenchymal Stem Cells for Treatment of CMV Infection After Hematopoietic Stem Cell Transplant
Brief Title: MSC for Treatment of CMV Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Academy Military Medical Science, China (Industry); Peking University People's Hospital (Other); Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSC-CMV-2014
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Stem Cell Transplantation, Hematopoietic; CMV Infection; Hematological Diseases
Keywords: CMV infection; Mesenchymal Stem Cells; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Cytomegalovirus Infections; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSCs (Experimental): MSCs will be used to treat refractory CMV infection or CMV-associated diseases. MSCs will be intravenously infused at a dose of 1×10^6 cells/kg. If anticipates do not attain the complete remission standards within 14d, a second course of the same treatment will be given.
  Interventions: Biological: MSCs

INTERVENTIONS:
Biological: MSCs

SUMMARY:
The purpose of this study is to evaluate the efficacy of mesenchymal stem cells (MSC) in the treatment of refractory cytomegalovirus (CMV) infection after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Viral infections are common complications after allo-HSCT. With wide use of HLA-mismatch, unrelated and cord blood donors as alternative sources of hematopoietic stem cells, and anti-thymocyte globulin (ATG) as the standard prophylaxis of graft versus host disease (GVHD) in HLA-mismatch and unrelated donor transplantation, allo-HSCT recipients are at increasing risk for viral infections.

Till now, CMV remains one of the most important viruses and causes of death in the recipients of allo-HSCT. Approximately 75% of CMV-seropositive recipients develop CMV reactivation, and 20-30% of these patients develop CMV disease without intervention. Ganciclovir is the first-line treatment of CMV diseases. However, bone marrow suppression, which is the main and common side effect, limits the utility of ganciclovir in allo-HSCT recipients. Besides, ganciclovir and other antiviral agents resistance has been reported up to 28%. Since it has been known that specific immune response to CMV is important to control reactivation, CMV-specific CTL has been used in prophylaxis and treatment of CMV viremia in several studies. However, the production of CTL requires time. Mesenchymal stem cells (MSC) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. In vivo experiment showed that MSCs have antimicrobial activity.

In this trial, we will use MSCs in the recipients with refractory CMV infections.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Refractory CMV infection or CMV-associated diseases
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants achieved complete remission of CMV infection | 1 year

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | up to 1 year
  Adverse Events include GVHD, primary underlying disease relapse and any other side effects. Side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Meisel R, Brockers S, Heseler K, Degistirici O, Bulle H, Woite C, Stuhlsatz S, Schwippert W, Jager M, Sorg R, Henschler R, Seissler J, Dilloo D, Daubener W. Human but not murine multipotent mesenchymal stromal cells exhibit broad-spectrum antimicrobial effector function mediated by indoleamine 2,3-dioxygenase. Leukemia. 2011 Apr;25(4):648-54. doi: 10.1038/leu.2010.310. Epub 2011 Jan 18. PMID 21242993
- [Background] Ljungman P, de la Camara R, Cordonnier C, Einsele H, Engelhard D, Reusser P, Styczynski J, Ward K; European Conference on Infections in Leukemia. Management of CMV, HHV-6, HHV-7 and Kaposi-sarcoma herpesvirus (HHV-8) infections in patients with hematological malignancies and after SCT. Bone Marrow Transplant. 2008 Aug;42(4):227-40. doi: 10.1038/bmt.2008.162. Epub 2008 Jun 30. PMID 18587440